CLINICAL TRIAL: NCT07246798
Title: The Effect of Preoperative Artificial Intelligence-Based Video Education on Anxiety and Anesthesia Preference in Patients Scheduled for Arthroscopic Lower Extremity Surgery
Brief Title: The Effect of Video Education on Anesthesia Choice
Status: Enrolling by invitation | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 25-MOBAEK-127
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia Education
Keywords: Test Anxiety Scale; Anesthesia; Patient Satisfaction; Patient Preference; Preoperative education; Arthroscopy
MeSH Terms: conditions — Patient Satisfaction; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The effect of AI-based video education on preoperative anxiety and anesthesia preference: Patients will watch an artificial intelligence-based preoperative video explaining anesthesia options and perioperative care. The Spielberger State Anxiety Inventory, satisfaction scale, and knowledge questionnaire will be applied before and after the video education. The impact of artificial intelligence-based video training on anesthesia preference will be evaluated.

SUMMARY:
This prospective single-group study aims to evaluate the effect of preoperative artificial intelligence-based video education on anxiety, anesthesia preference, satisfaction, and knowledge level in patients undergoing arthroscopic lower extremity surgery.

DETAILED DESCRIPTION:
Participants' demographic characteristics (age, gender, occupation, education level, income, marital status) will be recorded.

All patients will complete the Spielberger State Anxiety Inventory (STAI-I) before and after watching an AI-generated preoperative information video that explains anesthesia options and the perioperative process.

Their anesthesia preference, satisfaction, and knowledge level will also be assessed before and after the video.

The study aims to determine whether AI-based video education can reduce preoperative anxiety, alter anesthesia preference, and improve patient satisfaction and understanding.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective arthroscopic lower extremity surgery
* Able to understand the educational material
* Voluntarily agrees to participate and provides written informed consent

Exclusion Criteria:

* Mentally unable to provide valid responses
* Communication barriers or severe visual impairment
* Contraindication to regional or general anesthesia
* Illiteracy or inability to understand Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 65 years scheduled for elective arthroscopic lower extremity surgery at Tokat Gaziosmanpaşa University Faculty of Medicine Hospital, Department of Anesthesiology and Reanimation.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in anesthesia preference | Baseline (before the AI-assisted video information) and immediately after the AI-assisted video information, within the preoperative assessment period.
  The impact of artificial intelligence-based video training on anesthesia preference will be evaluated.
Change in Preoperative Anxiety Score (STAI-I) | Baseline (before the AI-assisted video information) and immediately after the AI-assisted video information, within the preoperative assessment period
  To evaluate whether AI-based video education reduces preoperative anxiety. The State Anxiety Inventory (STAI-I) is a validated self-report instrument consisting of 20 items assessing situational anxiety. Scores range from 20 to 80, with higher scores indicating greater anxiety. A higher score reflects a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data used to support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Researchers interested in accessing the data should contact the corresponding author via email with a brief description of their proposed use